CLINICAL TRIAL: NCT00012883
Title: Home Walking Exercise Training in Advanced Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRI 96-031
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-02

CONDITIONS: Heart Failure; Functional Status; Quality of Life
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other): Homewalking Exercise Program
  Interventions: Behavioral: Homewalking exercise program

INTERVENTIONS:
Behavioral: Homewalking exercise program

SUMMARY:
Heart failure is a major public health burden in the United States characterized by increased morbidity and mortality, and reduce exercise capacity with distressing symptoms of dyspnea and fatigue. Evaluating the effects of complementary intervention (such as exercise training) on functional status and QOL are clinically important and relevant to HF patients.

In the last decade, hospital-based and a home bicycle exercise programs for HF have been shown to improve peak oxygen consumption (VO2) and symptom scores, and restore autonomic balance. These programs may be costly for patients to perform. Improved peak VO2 may not necessarily translate into improved functional status and quality of life. To date, the effects of a home walking exercise program alone on functional status, QOL and autonomic tone has not been evaluated.

DETAILED DESCRIPTION:
Background:

Heart failure is a major public health burden in the United States characterized by increased morbidity and mortality, and reduce exercise capacity with distressing symptoms of dyspnea and fatigue. Evaluating the effects of complementary intervention (such as exercise training) on functional status and QOL are clinically important and relevant to HF patients.

In the last decade, hospital-based and a home bicycle exercise programs for HF have been shown to improve peak oxygen consumption (VO2) and symptom scores, and restore autonomic balance. These programs may be costly for patients to perform. Improved peak VO2 may not necessarily translate into improved functional status and quality of life. To date, the effects of a home walking exercise program alone on functional status, QOL and autonomic tone has not been evaluated.

Objectives:

The specific aim was to compare functional status (FS), quality of life (QOL) and autonomic tone in 2 groups of advanced HF patients (nurse-managed home walking exercise (HWE) group vs. control group).

Methods:

A randomized controlled trial comparing a 12-week nurse-managed progressive HWE protocol to usual activity was conducted in 79 HF patients (78[99%] male; mean age 62.6 � 10.6 years; EF 27 � 8.8%; 63 [80%] NYHA II, 15[20%] NYHA III-IV; HF duration 39.2 � 41.8 months) from a VA medical center and a university affiliated medical center. The 12- week HWE program is once a day, 5x a week and initiated at 10 minutes and progressively increases in duration and intensity up to 60 minutes. Pre- and post-study measures were FS (peak VO2 and ventilatory threshold via CPX, 6-minute walk test (6MWT) and a Heart Failure Functional Status Inventory (HFFSI)), QOL (Cardiac Quality of life Index (C-QLI), SF-36, and Dyspnea-Fatigue Index (DFI) with global rating of symptoms), and autonomic tone (norepinephrine (NE) and heart rate variability (HRV)). Intention-to-treat analysis with repeated measures ANOVA was used to identify group differences.

Status:

Completed.

ELIGIBILITY:
Inclusion Criteria:

Should have a stable heart failure in the past 3 months (Max Age is 80)

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Study Completion 2001-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teresita E. Corvera-Tindel, PhD RN MN, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (1):
- VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California, United States